CLINICAL TRIAL: NCT04273282
Title: The D3 Study: Drug Delivery vs Drops - A Prospective Clinical Study Evaluating Dexycu vs Prednisolone Acetate 1% in Controlling Post-operative Pain and Inflammation in Patients Undergoing Sequential Cataract Surgery
Brief Title: A Prospective Clinical Study Evaluating Dexycu vs Prednisolone Acetate 1%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1909 D3 EyePoint
Record Dates: First submitted 2019-12-18; First posted 2020-02-18 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — bromfenac; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: Each study subject will be randomized by a table in the possession of investigators to receive one of 2 treatment groups, either experimental or control in the first eye. The second eye will undergo cataract surgery approximately 2 weeks later and will be treated with the other treatment group:
  Dexycu Group:A total of 30 study subjects will have Dexycu intracameral dexamethasone placed in their scheduled surgical eye at the time of surgery and will receive 50 micrograms of intracameral moxifloxacin at the conclusion of the procedure. They will take Prolensa each day after surgery for 4 weeks.
  Control Group:A total of 30 study subjects will receive topical moxifloxacin 0.5% 4 times per day 1 day prior to surgery and for 10 days postoperatively, Prolensa every day 1 day prior to surgery and for 4 weeks postoperatively, and prednisolone acetate 1% four times per day starting at the conclusion of cataract surgery for 2 weeks and twice per day for 2 weeks in their scheduled surgical eye.
Who Masked: Participant
Masking Description: Only the participants will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexycu Group (Active Comparator): A total of 30 study subjects (30 eyes) will have Dexycu intracameral dexamethasone placed in their scheduled surgical eye at the time of surgery and will receive 50 micrograms of intracameral moxifloxacin at the conclusion of the procedure. They will take Prolensa qd after surgery for 4 weeks.
  Interventions: Drug: Dexycu intracameral dexamethasone
- Control Group (Active Comparator): A total of 30 study subjects (30 eyes) will receive topical moxifloxacin 0.5% qid 1 day prior to surgery and for ten days postoperatively, Prolensa qd 1 day prior to surgery and for 4 weeks postoperatively, and prednisolone acetate 1.0% qid starting at the conclusion of cataract surgery for 2 weeks and bid for 2 weeks in their scheduled surgical eye.
  Interventions: Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Dexycu intracameral dexamethasone — To evaluate the safety and ocular efficacy of Dexycu.
  Other Names: Moxifloxacin 0.5%; Prolensa
  Arms: Dexycu Group
Drug: Prednisolone Acetate — To evaluate the safety and ocular efficacy, and patient acceptance of post cataract surgery drug treatment regimen that minimizes topical medications.
  Arms: Control Group

SUMMARY:
This is a post-approval, open-label, randomized, self-controlled prospective clinical study to evaluate the safety and ocular efficacy of Dexycu in controlling postoperative ocular pain and inflammation associated with cataract surgery.

DETAILED DESCRIPTION:
On initial consultation, each study subject will be randomized by a table in the possession of investigators to receive one of two treatment groups, either experimental or control in the first eye. The second eye will undergo cataract surgery approximately 2 weeks later and will be treated with the other treatment group:

Dexycu Group: A total of 30 study subjects will have Dexycu intracameral dexamethasone placed in their scheduled surgical eye at the time of surgery and will receive 50 micrograms of intracameral moxifloxacin at the conclusion of the procedure. They will take Prolensa each day after surgery for 4 weeks.

Control Group: A total of 30 study subjects will receive topical moxifloxacin 0.5% four times per day 1 day prior to surgery and for ten days postoperatively, Prolensa every day 1 day prior to surgery and for 4 weeks postoperatively, and prednisolone acetate 1.0% four times per day starting at the conclusion of cataract surgery for 2 weeks and twice per day for 2 weeks in their scheduled surgical eye.

ELIGIBILITY:
Inclusion Criteria:

* A male or female in good general health, greater than 18 years of age at time of screening.
* Must be able to comprehend and willing to give informed consent.
* Woman of child-bearing potential must not be pregnant or lactating.
* Subject has availability, willingness, and sufficient cognitive awareness to comply with exam procedures and able to return for all scheduled study visits.
* Subject with cataract for which routine phacoemulsification extraction and implantation of an intraocular lens has been planned.
* Subject with an OCT of the macula in both eyes that demonstrates no significant pathology.

Exclusion Criteria:

* Subject with any signs of intraocular inflammation in either eye at screening.
* Subject with a known sensitivity to any of the study medications.
* Subject with only one eye with potentially good vision.
* Subject that has undergone prior intraocular surgery in the scheduled surgical eye within the last 6 months or laser surgery within three months prior to screening.
* Subject with pupil abnormalities.
* Subject with corneal abnormalities.
* Subject with a history of chronic/recurrent inflammatory eye disease in either eye.
* Subject with uncontrolled glaucoma.
* Subject expected to undergo surgical intervention and/or ocular laser treatment prior to or during the study period.
* Subject who requires use of systemic or ocular medications that may affect vision, ocular inflammation, or pain.
* Subject with an acute or chronic disease or illness that would increase risk or confound study results, e.g. autoimmune disease, etc.
* Subject with an uncontrolled systemic disease.
* Subject with poorly-controlled diabetes.
* Subject currently participating or has participated in another clinical trial within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Patient preference for medication protocol in 30 randomized subjects | Day 28
  Patient preference for medication protocol between the two eyes, as reported based on the question, "Thinking about your overall experience taking medications in each eye after surgery, which eye did you prefer? Questionnaire

SECONDARY OUTCOMES:
Subject evaluation of postop ocular pain in 30 randomized subjects | Day 28
  Study subject evaluation of post-op ocular pain.
Summed Ocular Inflammation Score in 30 randomized subjects | Day 28
  Summed Ocular Inflammation Score (sum of the mean anterior chamber cells and anterior flare score)
Medication cost in 30 randomized subjects | Day 28
  Cost of medications to the patient (patient-reported)

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — Research Insight LLC
Locations (2):
- United States (2):
  - Harvard Eye Associates, Laguna Hills, California
  - Ophthalmic Consultants of Long Island, Garden City, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hovanesian JA, Donnenfeld ED. Intracameral dexamethasone 9% vs prednisolone acetate 1% in controlling postoperative pain and inflammation in patients undergoing cataract surgery. J Cataract Refract Surg. 2022 Aug 1;48(8):906-911. doi: 10.1097/j.jcrs.0000000000000887. Epub 2022 Jan 18. PMID 35067660